CLINICAL TRIAL: NCT06818695
Title: Efficacy of Online Imaginal Exposure Therapy for Individuals With Anorexia Nervosa
Brief Title: Online Imaginal Exposure Therapy for Eating Disorders Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: North East London Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 162510
Record Dates: First submitted 2025-02-07; First posted 2025-02-10 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Anorexia Nervosa
Keywords: Intervention Study; Anorexia Nervosa; Imaginal Exposure; Waiting List Controls; Parallel Group Design
MeSH Terms: conditions — Anorexia Nervosa | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm (Experimental): Participants will receive imaginal exposure for Anorexia Nervosa
  Interventions: Other: Imaginal Exposure for Anorexia Nervosa
- Waitlist Control (Active Comparator): Participants in this arm will remain on the waitlist for the service and receive treatment as usual (TAU), which includes specialist nurse monitoring, occasional medical reviews, and dietetic support (depending on the individual's particular needs).
  Interventions: Other: Treatment as Usual (TAU)

INTERVENTIONS:
Other: Imaginal Exposure for Anorexia Nervosa — Imaginal exposure aims to use the power of imagining the fearful situation to heighten anxiety and by not engaging in imaginative restriction or other eating disorder behaviours, the individual, in theory, can habituate to the anxiety until it naturally subsides.
  Arms: Treatment Arm
Other: Treatment as Usual (TAU) — TAU includes specialist nurse monitoring, occasional medical reviews, and dietetic support (depending on the individual's particular needs)
  Arms: Waitlist Control

SUMMARY:
The goal of this clinical trial is to learn if an imaginal exposure intervention first conducted by Levinson and colleagues (2020) can produce similar promising results in individuals with anorexia on the waiting list of an NHS eating disorder service. The main question it aims to answer is:

1. How effective is Imaginal Exposure Therapy in reducing eating disorder symptoms and increasing weight in patients with AN?

   The secondary research questions are:
2. How effective is Imaginal Exposure Therapy in reducing anxiety and fear related outcomes around food and eating?
3. How effective is Imaginal Exposure Therapy in improving patients' general anxiety and depression symptoms?

Researchers will compare the results of individuals in the treatment condition to individual's in the control condition to explore the efficacy of the intervention on eating disorder and eating disorder fear symptomology, and body weight.

Participants in the intervention group will receive 4 sessions of online exposure therapy, and participants in the control group will remain on the waiting list with treatment as usual (primarily nurse monitoring).

DETAILED DESCRIPTION:
Study design type: The study will have a parallel group design. Approximately half of the participants will be randomised to receive our intervention, IE for AN. The other half will remain on the waitlist for the service and receive treatment as usual (TAU), which includes specialist nurse monitoring, occasional medical reviews, and dietetic support (depending on the individual's particular needs). This study design will allow us to directly assess the efficacy of the IE intervention, as compared to standard waiting list monitoring, on participants' weight and AN symptoms.

Sampling: Potential participants will be identified by the direct care team; any details not obtained through the study questionnaires will be obtained through digital medical records. The researchers will request information where needed through the direct care team. Participants will be recruited through the NELFT ED service post referral triage, while patients are on the waiting list. Participants will be the adults on the waiting list for receiving AN treatment at NELFT.

Procedure: Following informed consent, participation in the trial will last 5 weeks.

Week 1: All participants will, where possible, come to the service in-person to be weighed. All participants will complete a set of psychometric questionnaires during this appointment. The IE group will also complete the Eating Disorder Fear Interview (Levinson et al., 2019), administered in order to identify a fear to target in exposure therapy. If not possible to attend in-person, this primary appointment will be held on Zoom. All baseline appointments will be with a study coordinator.

Week 2: First online imaginal exposure. Week 3: Second online imaginal. Week 4: Third online imaginal exposure. Week 5: Fourth online imaginal exposure and participants will complete the final battery of online questionnaires. They will then come to the service in-person to be weighed again.

ELIGIBILITY:
Inclusion Criteria:

* Patients on the North East London Foundation Trust Eating Disorder waiting list.
* Patients who are over the age of 18 years old.
* Patients of all genders.
* Patients who have a primary diagnosis of Anorexia Nervosa.
* Patients who are willing and able to provide written informed consent.

Exclusion Criteria:

* Patients on the waiting list who are under the age of 18.
* Females who are pregnant, planning pregnancy or breastfeeding.
* Patients involved in concurrent research which is likely to interfere with the imaginal exposure intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Eating Disorder Examination Questionnaire | From initial interview till the end of treatment after 5 weeks
  A 28-item questionnaire aiming to assess the characteristics, range, frequency and severity of behaviours associated with clinical eating disorders such as Anorexia Nervosa, Bulimia Nervosa, Binge Eating Disorder and OSFED. It consists of 4 subscales: Restraint, Eating Concern, Shape Concern and Weight Concern and overall global score. Higher scores are indicative of more severe eating difficulties and the scale is used as an assessment and diagnostic tool.
Body Mass Index | From initial session until the end of intervention at 5 weeks
  BMI is a measure using an individual's tissue mass (weight) and height to determine body mass index, which is categorised into the following: Underweight (under 18.5 kg/m2), Normal Weight (18.5-24.9) Overweight (25-29.9) and Obese (30 or more).

SECONDARY OUTCOMES:
Fear of Food Measure (FOFM) | From initial session to the end of the intervention at 5 weeks
  Designed by Levinson et al., specifically to assess improvement in Eating Related Anxiety over the course of Imagined Exposure Therapy. It consists of 3 subscales: Anxiety about Eating, Food Avoidance Behaviours, and Feared Concerns.
Eating Disorder Fears Interview (EFI) | From initial session to the end of intervention at 5 weeks
  Designed by Levinson et al., the EFI is a semi-structured interview consisting of 31 items designed to assess common ED fears such as food, weight gain and consequences of weight gain (judgement). This interview can also be used in tandem with Eating Disorder clinical assessment interviews to attain a more in depth understanding of treatment aims and goals.
Eating Disorder Fears Questionnaire (EFQ) | From initial session to the end of intervention at 5 weeks
  Designed by Levinson et al., the EFQ is a 30 item self-report measure designed to assess common ED fears such as gaining weight, consequences of weight gain, and eating in public.
Penn State Worry Questionnaire (PSWQ) | From initial session to end of intervention at 5 weeks.
  A 16 Item Questionnaire assessing traits of worrying in adults. The scale measures three dimensions of worrying: excessive, generality and uncontrollable.
Beck Depression Inventory II (BDI-II) | From the initial session to the end of the intervention at 5 weeks.
  The BDI-II is a 21 item self report inventory measuring severity of depression in adolescents and adults.

CONTACTS AND LOCATIONS:
Overall Officials: Lucy Serpell, Principal Investigator — University College, London
Locations (1):
- North East London Foundation Trust Eating Disorder Service, London, Barking, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levinson CA, Christian C, Ram SS, Vanzhula I, Brosof LC, Michelson LP, Williams BM. Eating disorder symptoms and core eating disorder fears decrease during online imaginal exposure therapy for eating disorders. J Affect Disord. 2020 Nov 1;276:585-591. doi: 10.1016/j.jad.2020.07.075. Epub 2020 Jul 21. PMID 32794449